CLINICAL TRIAL: NCT07016763
Title: Combination of Oral Supplement With Fatty Acids, Vitamin B6, Perilla, and Liquorice With Nasal Steroids for the Treatment of Allergic Rhinitis: a Multicentre, Single-blinded, Randomized Controlled Trial
Brief Title: Combination of Oral Supplement With Fatty Acids, Vitamin B6, Perilla, and Liquorice With Nasal Steroids for the Treatment of Allergic Rhinitis
Acronym: LT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Isola Tiberina - Gemelli Isola Hospital, Rome, Italy (Other)
Responsible Party: Principal Investigator, Pietro De Luca, MD, Consultant, Isola Tiberina - Gemelli Isola Hospital, Rome, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/2025
Record Dates: First submitted 2025-05-20; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; intranasal corticosteroids; rhinosinusitis; fatty acid
MeSH Terms: conditions — Rhinitis, Allergic; Rhinosinusitis | interventions — Fatty Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intranasal corticosteroids + oral fatty acids
  Interventions: Dietary Supplement: Oral fatty acid
- Control group (Active Comparator): Intranasal corticosteroids alone
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)

INTERVENTIONS:
Dietary Supplement: Oral fatty acid — Intervention therapy (treatment group) daily treated for 90 consecutive days by INCs (mometasone furoate; 1 puff in each nostril, twice a day) and oral supplementation of FAs (550 mg/tablet), vitamin B6 (0.21 mg/tablet), perilla frutescens (20 mg/tablet) and liquorice (200/mg/tablet) (2 tablets a day with meals)
  Arms: Intervention Group
Drug: Mometasone Furoate Nasal Spray (MFNS) — Standard therapy (control group) daily treated for 90 consecutive days by INCs (mometasone furoate; 1 puff in each nostril, twice a day) only
  Arms: Control group

SUMMARY:
Previous studies on the association between the development of allergic diseases and diet indicate the involvement of dietary fatty acids (FA) in the acceleration and/or inhibition of allergic diseases. Edible oils contain various FAs, but their composition depends on the materials from which they are extracted. FAs are characterised by the presence or absence of a carbon double bond in their structure; saturated FAs (palmitic acid, stearic acid, etc.) have no carbon double bond, while unsaturated FAs contain at least one carbon double bond. Among the unsaturated FAs, omega-3 FAs (such as alpha-linolenic acid [ALA], eicosapentaenoic acid [EPA] and docosahexaenoic acid [DHA]) and omega-6 FAs (such as linoleic acid [LA] and arachidonic acid [ARA]) are classified as essential FAs. Various types of bioactivity of dietary essential FAs have been reported in health and disease studies, including immunity, allergy and inflammation. Human studies, for example, have shown an association between the quality of dietary FAs and the incidence of allergic diseases.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;
* confirmed diagnosis of AR already treated with scarce or absent results by general practitioners

Exclusion Criteria:

* pregnancy or breastfeeding;
* concomitant asthma without stable control;
* chronic obstructive and restrictive lung disease;
* autoimmune and collagen diseases;
* acute sinusitis, nasal or upper respiratory tract infections in acute phase;
* cardiovascular, hepatic, or renal disease;
* other poorly controlled serious or chronic diseases;
* taking medications that may affect the immune response;
* previous nasal surgery;
* immunotherapy in the 3 years prior to enrolment, or the ones who planned to receive immunotherapy;
* patients who did not sign the informed consent for;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic evaluation | From the enrolment (T0, baseline, diagnosis) to T1 (90 days after the diagnosis and treatment start)
  Endoscopic evaluation of the nose using the Lund-Kennedy (LK) score.THe LK scoring system is based on the degree of polyps, discharge and edema in each nostril.
Symptoms and quality of life evaluation, VAS | From the enrolment (T0, baseline, diagnosis) to T1 (90 days after the diagnosis and treatment start)
  Symptoms and quality of life evaluation using the Visual Analog Scale (VAS, range 0-10; >5= uncontrolled disease)
Symptoms and quality of life evaluation, MiniRQoLQ | From the enrolment (T0, baseline, diagnosis) to T1 (90 days after the diagnosis and treatment start)
  Symptoms and quality of life evaluation using the Visual Analog Scale (VAS, range 0-10; >5= uncontrolled disease) and Mini Rhinoconjuctivitis Quality of Life Questionnaire (MiniRQoLQ, which utilizes a 7-point scale for each of its 14 questions, ranging from 0 (not impaired at all) to 6 (severely impaired), ranging 0-84).

CONTACTS AND LOCATIONS:
Locations (1):
- Isola Tiberina Hospital, Rome, Italy, Italy